CLINICAL TRIAL: NCT01154998
Title: Case-Control Study of Fibrotic Interstitial Lung Disease and it's Association With Cardiac Disease or Cardiac Intervention.
Brief Title: Case-Control Study of Fibrotic Interstitial Lung Disease (ILD) and Cardiac Disease / Interventions.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: St George's Healthcare NHS Trust (Other)
Responsible Party: Dr Felix Chua, St George's Healthcare NHS Trust
Other Study IDs: 10/H1102/46
Record Dates: First submitted 2010-06-30; First posted 2010-07-01 (Estimated); Last update posted 2010-07-01 (Estimated); Status verified 2010-06

CONDITIONS: Idiopathic Pulmonary Fibrosis; Interstitial Pneumonia
Keywords: non-specific interstitial pneumonia
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases
- Controls

SUMMARY:
There is a rare condition causing scarring of the lungs termed interstitial lung disease. This comprises a group of conditions which can be divided into separate diseases. The aim of this study is compare a group of patients (the cases) with 2 types of this disease (fibrotic non-specific interstitial pneumonia (NSIP) and idiopathic pulmonary fibrosis (IPF)) with patients without the disease. The study will look at the 2 groups and their exposures to factors such as medications, smoking, previous jobs, previous medical problems and specifically heart disease and any operations or procedures involving the heart. There have been previous studies showing a link between heart disease and scarring of the lungs. This study will look at whether this association is stronger in one or the other type of lung scarring diseases.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic fibrotic lung disease

Exclusion Criteria:

* non idiopathic fibrotic lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases - patients with IPF or UIP. Controls - hospital clinic attenders.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-01 (Estimated); Study Completion 2011-04 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- St George's Hospital, London, London, United Kingdom